CLINICAL TRIAL: NCT03157557
Title: Multidisciplinary Lifestyle-enhancing Treatment for Long-term Severe Mentally Ill Inpatients: Sheltered Housing
Brief Title: Multidisciplinary Lifestyle-enhancing Treatment for People With Severe Mental Illness in Sheltered Housing Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GGZ Centraal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL61552.075.17
Record Dates: First submitted 2017-05-08; First posted 2017-05-17 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Lifestyle; Mental Disorders, Severe
Keywords: Treatment; Sheltered Housing
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle treatment (Experimental): Lifestyle treatment
  Interventions: Behavioral: Lifestyle treatment
- Treatment as Usual (No Intervention): Treatment as Usual

INTERVENTIONS:
Behavioral: Lifestyle treatment — Lifestyle treatment
  Arms: Lifestyle treatment

SUMMARY:
Introduction and rationale:

Unhealthy eating habits and lack of physical activity are risk factors for many diseases (including metabolic syndrome) and contribute to a shortened lifespan of 15-30 years in people with severe mental illness (SMI). Literature, mainly including short-term hospitalized or outpatients, show strong positive effects of activation on both physical and mental health. However, studies in long-term care are limited. In recent years, implementation of a lifestyle enhancing treatment intervention in clinical settings in "GGz Centraal" has demonstrated to be effective. The question is whether this kind of lifestyle intervention in sheltered housing is applicable and effective.

Objectives:

This research aims to develop an appropriate lifestyle intervention for patients living in sheltered housing services of GGz Centraal, based on input of patients and directly involved. Does applying this lifestyle treatment result in a positive effect in health and quality of life of patients and what is the influence of contextual factors, personal- and disease characteristics?

Study design:

In this intervention study, we use an experimental design. Municipal locations are paired based on the number of participants to generate equal cluster sizes. These paired clusters are randomly allocated to the control or intervention arm by means of a random number generator by an independent person (not involved in this project). At the start of the lifestyle treatment patients in the experimental and control group are invited to participate in the baseline screening. After twelve months, following a post-test on all outcome measures.

Treatment intervention:

The intervention in this study consists of formulating a lifestyle intervention, by patients and directly involved, aimed at enhancing a more active and healthier lifestyle . After formulation of the plan (based on psycho education, nutrition and physical activity), it wil be executed for a twelve month period.

Hypothesis:

Hypotheses is that lifestyle enhancing treatment is associated with improved metabolic health, quality of life and reduced use of medication. Furthermore we expect that movement disorders and disease severity will be negative related in becoming more active.

DETAILED DESCRIPTION:
Sample size calculation:

To calculate the sample size we use the effect size on decrease in waist circumference in the previous intervention study (d =0.51) and the same analysis (multiple regression with correction for baseline value's on age, diagnosis and disease severity). To be able to detect the same effect in the current study with a minimum 80% power as a benchmark for a fair test and a significant level of 95% (α = 0.05), a minimum sample of 124 people is required (2 groups of 62). Taking into account a response rate of 73% from the first measurement a sample size of 168 patients is required.

Analyses:

We use multilevel regression to analyze the intervention effect. Possible clustering of data within the residential locations (and thus care teams) is taken into account by using a two-level structure with the first level residential location and the patients as the second. The intervention variable is set as an independent variable against difference scores of outcome variables (T2 minus T1) and corrected for the baseline value of the outcome to prevent regression to the centre. As we are unable to randomize patients individually in the current configuration on personal and disease characteristics (gender, age, diagnosis, disease severity at the start of intervention), these factors will be corrected for in the analyses if they differ significantly(p<0.05) between intervention and control group, analysed using independent t-tests and chi-squared tests. Characteristics that differ significantly will be included as covariates in the analysis described above. Multicollinearity will be checked with correlation coefficients and collinearity statistics (tolerance and Variance Inflation Factors (VIF) values).

Missing data:

Patients who are hospitalized for more than two months will be excluded from analyses.

If baseline or follow-up data are missing for two or more measures on physical or psychiatric health, patients are excluded from the analysis as insufficient difference scores can be calculated. Patients lacking difference scores on one outcome variable, are excluded from the analysis of that particular variable.

ELIGIBILITY:
Inclusion Criteria:

* Severe Mentally Ill patients,
* living in Sheltered Housing facilities

Exclusion Criteria:

* Incapacitated patients,
* without informed consent from their legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-05-17 (Actual)

PRIMARY OUTCOMES:
Metabolic Health: Waist circumference | 12 months
  measured halfway between the iliac crest and lowest rib in standing position

SECONDARY OUTCOMES:
Metabolic Health: weight | 12 months
  weight measured to the nearest 0.1kg
Metabolic Health: blood pressure | 12 months
  measured systolic and diastolic blood pressure (mmHg)
Metabolic Health:Lipids | 12 months
  values in blood sample
Metabolic Health:Fasting glucose | 12 months
  values in blood sample
Metabolic health: HbA1c | 12 months
  values in blood sample
Sedentary behaviour & physical activity | 12 months
  measured 5 consecutive days with an accelerometer (ActiGraph GT3X+
Quality of Life EuroQol 5D | 12 months
  measured by the EuroQol 5D (EQ-5D)
Quality of Life WHOQoL | 12 months
  measured by the WHOQoL-Bref
Psychopathology BPRS-E | 12 months
  Psychopathology / illness severity measured by the BPRS-E
Implementation fidelity | At follow-up (12 months)
  A proxy for implementation fidelity using the 'descriptive norm' item of the Measurement Instrument for Determinants of Innovations

CONTACTS AND LOCATIONS:
Overall Officials: Peter N van Harten, Prof. Dr., Study Director — GGZ Centraal
Locations (1):
- Veldwijk, Ermelo, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acil AA, Dogan S, Dogan O. The effects of physical exercises to mental state and quality of life in patients with schizophrenia. J Psychiatr Ment Health Nurs. 2008 Dec;15(10):808-15. doi: 10.1111/j.1365-2850.2008.01317.x. PMID 19012672
- [Background] Aleman A, Hijman R, de Haan EH, Kahn RS. Memory impairment in schizophrenia: a meta-analysis. Am J Psychiatry. 1999 Sep;156(9):1358-66. doi: 10.1176/ajp.156.9.1358. PMID 10484945
- [Background] Andreasen NC, Carpenter WT Jr, Kane JM, Lasser RA, Marder SR, Weinberger DR. Remission in schizophrenia: proposed criteria and rationale for consensus. Am J Psychiatry. 2005 Mar;162(3):441-9. doi: 10.1176/appi.ajp.162.3.441. PMID 15741458
- [Background] Bassett DR Jr, Cureton AL, Ainsworth BE. Measurement of daily walking distance-questionnaire versus pedometer. Med Sci Sports Exerc. 2000 May;32(5):1018-23. doi: 10.1097/00005768-200005000-00021. PMID 10795795
- [Background] Bech P, Larsen JK, Andersen J. The BPRS: psychometric developments. Psychopharmacol Bull. 1988;24(1):118-21. No abstract available. PMID 3387515
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Callaghan P. Exercise: a neglected intervention in mental health care? J Psychiatr Ment Health Nurs. 2004 Aug;11(4):476-83. doi: 10.1111/j.1365-2850.2004.00751.x. PMID 15255923
- [Background] Daumit GL, Goldberg RW, Anthony C, Dickerson F, Brown CH, Kreyenbuhl J, Wohlheiter K, Dixon LB. Physical activity patterns in adults with severe mental illness. J Nerv Ment Dis. 2005 Oct;193(10):641-6. doi: 10.1097/01.nmd.0000180737.85895.60. PMID 16208158
- [Background] Delespaul PH; de consensusgroep EPA. [Consensus regarding the definition of persons with severe mental illness and the number of such persons in the Netherlands]. Tijdschr Psychiatr. 2013;55(6):427-38. Dutch. PMID 23864410
- [Background] Dingemans PM, Linszen DH, Lenior ME, Smeets RM. Component structure of the expanded Brief Psychiatric Rating Scale (BPRS-E). Psychopharmacology (Berl). 1995 Dec;122(3):263-7. doi: 10.1007/BF02246547. PMID 8748395
- [Background] Docx L, Sabbe BG, Koning J, Mentzel TQ, van Harten PN, Morrens M. [Instrumental registration of psychomotor symptoms in schizophrenia: has the time come to use the technique in clinical practice?]. Tijdschr Psychiatr. 2015;57(2):148-53. Dutch. PMID 25669955
- [Background] Farnam CR, Zipple AM, Tyrrell W, Chittinanda P. Health status risk factors of people with severe and persistent mental illness. J Psychosoc Nurs Ment Health Serv. 1999 Jun;37(6):16-21. doi: 10.3928/0279-3695-19990601-15. PMID 10382153
- [Background] Foussias G, Remington G. Negative symptoms in schizophrenia: avolition and Occam's razor. Schizophr Bull. 2010 Mar;36(2):359-69. doi: 10.1093/schbul/sbn094. Epub 2008 Jul 21. PMID 18644851
- [Background] Gerlach J, Korsgaard S, Clemmesen P, Lauersen AM, Magelund G, Noring U, Povlsen UJ, Bech P, Casey DE. The St. Hans Rating Scale for extrapyramidal syndromes: reliability and validity. Acta Psychiatr Scand. 1993 Apr;87(4):244-52. doi: 10.1111/j.1600-0447.1993.tb03366.x. PMID 8098178
- [Background] Hafkenscheid A. Psychometric evaluation of the Nurses Observation Scale for Inpatient Evaluation in The Netherlands. Acta Psychiatr Scand. 1991 Jan;83(1):46-52. doi: 10.1111/j.1600-0447.1991.tb05510.x. PMID 2011956
- [Background] Kane I, Lee H, Sereika S, Brar J. Feasibility of pedometers for adults with schizophrenia: pilot study. J Psychiatr Ment Health Nurs. 2012 Feb;19(1):8-14. doi: 10.1111/j.1365-2850.2011.01747.x. Epub 2011 May 25. PMID 22070156
- [Background] Killaspy H, White S, Wright C, Taylor TL, Turton P, Kallert T, Schuster M, Cervilla JA, Brangier P, Raboch J, Kalisova L, Onchev G, Alexiev S, Mezzina R, Ridente P, Wiersma D, Visser E, Kiejna A, Piotrowski P, Ploumpidis D, Gonidakis F, Caldas-de-Almeida JM, Cardoso G, King M. Quality of longer term mental health facilities in Europe: validation of the quality indicator for rehabilitative care against service users' views. PLoS One. 2012;7(6):e38070. doi: 10.1371/journal.pone.0038070. Epub 2012 Jun 4. PMID 22675508
- [Background] Kozey-Keadle S, Libertine A, Lyden K, Staudenmayer J, Freedson PS. Validation of wearable monitors for assessing sedentary behavior. Med Sci Sports Exerc. 2011 Aug;43(8):1561-7. doi: 10.1249/MSS.0b013e31820ce174. PMID 21233777
- [Background] Kruisdijk F, Deenik J, Tenback D, Tak E, Beekman AJ, van Harten P, Hopman-Rock M, Hendriksen I. Accelerometer-measured sedentary behaviour and physical activity of inpatients with severe mental illness. Psychiatry Res. 2017 Aug;254:67-74. doi: 10.1016/j.psychres.2017.04.035. Epub 2017 Apr 22. PMID 28456024
- [Background] Mas-Exposito L, Amador-Campos JA, Gomez-Benito J, Lalucat-Jo L; Research Group on Severe Mental Disorder. The World Health Organization Quality of Life Scale Brief Version: a validation study in patients with schizophrenia. Qual Life Res. 2011 Sep;20(7):1079-89. doi: 10.1007/s11136-011-9847-1. Epub 2011 Feb 3. PMID 21290191
- [Background] Millier A, Schmidt U, Angermeyer MC, Chauhan D, Murthy V, Toumi M, Cadi-Soussi N. Humanistic burden in schizophrenia: a literature review. J Psychiatr Res. 2014 Jul;54:85-93. doi: 10.1016/j.jpsychires.2014.03.021. Epub 2014 Apr 4. PMID 24795289
- [Background] Ozemek C, Kirschner MM, Wilkerson BS, Byun W, Kaminsky LA. Intermonitor reliability of the GT3X+ accelerometer at hip, wrist and ankle sites during activities of daily living. Physiol Meas. 2014 Feb;35(2):129-38. doi: 10.1088/0967-3334/35/2/129. Epub 2014 Jan 7. PMID 24399138
- [Background] Rossler W, Salize HJ, van Os J, Riecher-Rossler A. Size of burden of schizophrenia and psychotic disorders. Eur Neuropsychopharmacol. 2005 Aug;15(4):399-409. doi: 10.1016/j.euroneuro.2005.04.009. PMID 15925493
- [Background] Sallis JF, Saelens BE. Assessment of physical activity by self-report: status, limitations, and future directions. Res Q Exerc Sport. 2000 Jun;71(2 Suppl):S1-14. No abstract available. PMID 10925819
- [Background] Santos-Lozano A, Santin-Medeiros F, Cardon G, Torres-Luque G, Bailon R, Bergmeir C, Ruiz JR, Lucia A, Garatachea N. Actigraph GT3X: validation and determination of physical activity intensity cut points. Int J Sports Med. 2013 Nov;34(11):975-82. doi: 10.1055/s-0033-1337945. Epub 2013 May 22. PMID 23700330
- [Background] Sasaki JE, John D, Freedson PS. Validation and comparison of ActiGraph activity monitors. J Sci Med Sport. 2011 Sep;14(5):411-6. doi: 10.1016/j.jsams.2011.04.003. Epub 2011 May 25. PMID 21616714
- [Background] Soundy A, Roskell C, Stubbs B, Vancampfort D. Selection, use and psychometric properties of physical activity measures to assess individuals with severe mental illness: a narrative synthesis. Arch Psychiatr Nurs. 2014 Apr;28(2):135-51. doi: 10.1016/j.apnu.2013.12.002. Epub 2013 Dec 19. PMID 24673789
- [Background] Stanton R, Happell B. Exercise for mental illness: a systematic review of inpatient studies. Int J Ment Health Nurs. 2014 Jun;23(3):232-42. doi: 10.1111/inm.12045. Epub 2013 Sep 30. PMID 24119136
- [Background] Stubbs B, Firth J, Berry A, Schuch FB, Rosenbaum S, Gaughran F, Veronesse N, Williams J, Craig T, Yung AR, Vancampfort D. How much physical activity do people with schizophrenia engage in? A systematic review, comparative meta-analysis and meta-regression. Schizophr Res. 2016 Oct;176(2-3):431-440. doi: 10.1016/j.schres.2016.05.017. Epub 2016 Jun 1. PMID 27261419
- [Background] Tenback DE, van Kessel F, Jessurun J, Pijl YJ, Heerdink ER, van Harten PN. [Risk factors for inactivity in patients in long-term care with severe mental illness]. Tijdschr Psychiatr. 2013;55(2):83-91. Dutch. PMID 23408360
- [Background] Thornicroft G, Tansella M. The balanced care model for global mental health. Psychol Med. 2013 Apr;43(4):849-63. doi: 10.1017/S0033291712001420. Epub 2012 Jul 11. PMID 22785067
- [Background] van Os J, Kapur S. Schizophrenia. Lancet. 2009 Aug 22;374(9690):635-45. doi: 10.1016/S0140-6736(09)60995-8. PMID 19700006
- [Background] Vancampfort D, Probst M, Scheewe T, Maurissen K, Sweers K, Knapen J, De Hert M. Lack of physical activity during leisure time contributes to an impaired health related quality of life in patients with schizophrenia. Schizophr Res. 2011 Jul;129(2-3):122-7. doi: 10.1016/j.schres.2011.03.018. Epub 2011 Apr 14. PMID 21493044
- [Background] Vancampfort D, Rosenbaum S, Schuch F, Ward PB, Richards J, Mugisha J, Probst M, Stubbs B. Cardiorespiratory Fitness in Severe Mental Illness: A Systematic Review and Meta-analysis. Sports Med. 2017 Feb;47(2):343-352. doi: 10.1007/s40279-016-0574-1. PMID 27299747
- [Background] Vancampfort D, Stubbs B, Mitchell AJ, De Hert M, Wampers M, Ward PB, Rosenbaum S, Correll CU. Risk of metabolic syndrome and its components in people with schizophrenia and related psychotic disorders, bipolar disorder and major depressive disorder: a systematic review and meta-analysis. World Psychiatry. 2015 Oct;14(3):339-47. doi: 10.1002/wps.20252. PMID 26407790
- [Background] Walker ER, McGee RE, Druss BG. Mortality in mental disorders and global disease burden implications: a systematic review and meta-analysis. JAMA Psychiatry. 2015 Apr;72(4):334-41. doi: 10.1001/jamapsychiatry.2014.2502. PMID 25671328
- [Derived] Smit MMC, Waal E, Tenback DE, Deenik J. Evaluating the implementation of a multidisciplinary lifestyle intervention for people with severe mental illness in sheltered housing: effectiveness-implementation hybrid randomised controlled trial. BJPsych Open. 2022 Nov 22;8(6):e201. doi: 10.1192/bjo.2022.600. PMID 36412504